CLINICAL TRIAL: NCT03438890
Title: Randomized Comparison of Laparoscopic LEns Defogging Using Anti-fog Solution, waRm Saline, and Chlorhexidine Solution (CLEAR)
Brief Title: Laparoscopic Lens Defogging Using Anti-fog Solution, waRm Saline, and Chlorhexidine Solution
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-03-005
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation information was hidden from the participants and outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Warm saline group (Experimental): In subjects allocated to the warm saline group, a thermos flask, which was filled with heated sterile water, was used. A 1000 ml bottle of sterile water was heated to 60 ˚C in a stove for an hour at minimum. Just before introducing into the abdominal cavity, the laparoscope was placed into the thermos flask for 30 seconds at minimum . After each incidence of laparoscopic lens fogging (LLF), the scope was briefly inserted into the thermos flask about 10 seconds, and was then wrapped gauze around the lens before abdominal reinsertion.
  Interventions: Device: Warm saline
- anti-fog agent group (Experimental): In the anti-fog agent group, Ultra-Stop TM (Sigmaphrarm, Vienna, Austria), which is a commercial anti-fogging solution containing alcohol, surfactant, and water for medical optical devices, was used. Wiping the lens with gauze soaked in Ultra-Stop TM and allowing the surfactant to act for 5 seconds, the laparoscope was introduced into the abdominal cavity. After each laparoscopic lens fogging (LLF), the scope was removed from the abdomen and cleaned using the same corresponding method.
  Interventions: Device: anti-fog agent
- chlorhexidine group (Experimental): In the chlorhexidine group, the lens was wiped with gauze soaked in 4% chlorhexidine detergent solution (Firson, Cheonan, Korea) for 5 seconds before introducing into the abdominal cavity, and chlorhexidine was reapplied on the lens at the occurrence of laparoscopic lens fogging (LLF).
  Interventions: Device: chlorhexidine
- control group (No Intervention): In the control group, the lens was not wiped gauze or applied any solution before use of the laparoscope. When occurred the event of each laparoscopic lens fogging (LLF) that splatter of irrigation fluid, blood, and body fluids affected visual clearance, the laparoscopic lens was manually rubbed with clean gauze by a scrub nurse.

INTERVENTIONS:
Device: Warm saline — In subjects allocated to the warm saline group, a thermos flask, which was filled with heated sterile water, was used. A 1000 ml bottle of sterile water was heated to 60 ˚C in a stove for an hour at minimum. Just before introducing into the abdominal cavity, the laparoscope was placed into the thermos flask for 30 seconds at minimum . After each incidence of laparoscopic lens fogging (LLF), the scope was briefly inserted into the thermos flask about 10 seconds, and was then wrapped gauze around the lens before abdominal reinsertion.
  Arms: Warm saline group
Device: anti-fog agent — In the anti-fog agent group, Ultra-Stop TM (Sigmaphrarm, Vienna, Austria), which is a commercial anti-fogging solution containing alcohol, surfactant, and water for medical optical devices, was used. Wiping the lens with gauze soaked in Ultra-Stop TM and allowing the surfactant to act for 5 seconds, the laparoscope was introduced into the abdominal cavity. After each laparoscopic lens fogging (LLF), the scope was removed from the abdomen and cleaned using the same corresponding method.
  Arms: anti-fog agent group
Device: chlorhexidine — In the chlorhexidine group, the lens was wiped with gauze soaked in 4% chlorhexidine detergent solution (Firson, Cheonan, Korea) for 5 seconds before introducing into the abdominal cavity, and chlorhexidine was reapplied on the lens at the occurrence of laparoscopic lens fogging (LLF).
  Arms: chlorhexidine group

SUMMARY:
The aim of this study is to compare three popular methods of minimizing or reducing laparoscopic lens fogging (LLF) by heating lens using warm saline, applying anti-fog agent to lens, and rubbing lens with chlorhexidine in laparoscopic gynecologic surgery.

DETAILED DESCRIPTION:
The physiology behind laparoscopic lens fogging (LLF) is well understood based on meticulous experiments outlining the role of temperature and humidity. Despite many efforts, including uses of warm saline, various anti-fog agents, chlorhexidine, betadine, and rubbing the lens on serosal surfaces, to reduce LLF, there remains no consensus as to which method is superior to prevent LLF. Furthermore, most previous studies were experimental trials conducted in a simulation model or a non-human in vivo model or an expert's commentary based on their clinical experiences , and there was no randomized controlled trial focusing LLF in human model. Therefore, this randomized trial aimed to compare three popular methods of minimizing or reducing LLF by heating lens using warm saline, applying anti-fog agent to lens, and rubbing lens with chlorhexidine in laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* the absence of pregnancy at the time of surgery

Exclusion Criteria:

* allergy to chlorhexidine or anti-fog solution
* anticipating cases of abrupt change in intra-abdominal humidity such as hemoperitoneum and profuse ascites
* extremely short or long operative time (<20 min or > 180 min) affecting the frequency of LLF
* unavailability of the surgical recording equipment for laparoscopic procedure.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
the severity of LLF during the first 3-min operation | At the time of surgery
  The severity of LLF was rated on a scale of 0 (the clearest) to 10 (the foggiest).

SECONDARY OUTCOMES:
the severity of LLF occurred during the remaining operative time except the first 3-min | At the time of surgery
  The severity of LLF was rated on a scale of 0 (the clearest) to 10 (the foggiest).
the number of lens cleansing | At the time of surgery
  We will assess the number of lens cleansing at the time of surgery.
total time to spend for lens cleaning | At the time of surgery
  We will assess the total time to spend for lens cleansing at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No